CLINICAL TRIAL: NCT04164498
Title: Noise in Critical Care Units.Impact on Critically Ill Patients and Healthcare Personnel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Fakher, Assistant professor(lecturer), Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-15-2019
Record Dates: First submitted 2019-11-07; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Noise; Adverse Effect
Keywords: Noise ICU; delirium; depression; burnout; music
MeSH Terms: conditions — Delirium; Depression; Burnout, Psychological | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music exposure (Experimental): will be exposed to music to investigate effects on preventing noise Adverse effects
  Interventions: Other: music
- Control (No Intervention): no exposure to music

INTERVENTIONS:
Other: music — exposure to music to investigate its effects on reducing noise adverse effects
  Arms: Music exposure

SUMMARY:
Study noise level in the ICU and its effect on both patients and healthcare personnel.

Use music and study same effects on same patients and healthcare personnel.

DETAILED DESCRIPTION:
Level of noise is measured and investigate its effects on delirium prevalence. sleep quality score. hemodynamics of patients.

burnout and depressive symptoms of healthcare personnel

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to ICU fully conscious and can answer the questionnaires of the study

Exclusion Criteria:

* confused patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-09 (Estimated); Primary Completion 2019-12-05 (Estimated); Study Completion 2019-12-05 (Estimated)

PRIMARY OUTCOMES:
sleep quality: Richard Campbell sleep questionnaire | 1 month
  Richard Campbell sleep questionnaire will be used A modified 6 question questionnaire each question from 0 to 100
delirium | in hospital up to 2 months
  Confusion Assessment Method flow sheet in ICU (CAM -ICU too)l will be used 4 questions flow sheet
Burnout syndrome | 1 month
  Occurrence of burnout syndrome in healthcare personnel
Depression symptoms | 1 month
  Occurrence of depression symptoms in healthcare personnel assessed by becks tool

SECONDARY OUTCOMES:
length of stay in icu | in hospital 1 year
  Length of patient stay in the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Amin Fakher, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No